CLINICAL TRIAL: NCT05430542
Title: Different Variations of Intra-familial Body Mass Index Subjected to COVID-19 Lockdown
Brief Title: Age-related Post-lockdown BMI Variations
Acronym: COVIDLOCKMET01
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, MD, University of Bari
Other Study IDs: COVID-LOCKDOWN MET 01
Record Dates: First submitted 2022-06-23; First posted 2022-06-24 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Metabolic Syndrome; Overweight and Obesity
Keywords: Body mass index; COVID-19; Diet; Lockdown; Overweight and Obesity; Physical activity; Sedentary behavior
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; COVID-19; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 lockdown has represented an unedited model of increased metabolic risk in all age groups, due to negative changes in dietary habits, physical activity, lifestyle. These effects have been generally explored at a population level in distinct age groups. Potential intra-familial, specific effects in adults and children sharing the same socio-economic, cultural level and living habits have been scarcely explored. The investigators aimed to extend the previous observations concerning anthropometric data at the intra-familial level. In particular, The investigators prospectively characterized the variations in lifestyle habits and related outcomes over a 2 two months COVID-19 lockdown period, exploring both parents and their children. A cohort of 149 couple parent/children were prospectively enrolled. By a validated questionnaire The investigators explored changes of Body Mass Index (BMI) and individual lifestyle during a 2-month lockdown.

DETAILED DESCRIPTION:
The COVID-19 lockdown has represented an unedited model of increased metabolic risk in all age groups, due to negative changes in dietary habits, physical activity, lifestyle. These effects have been generally explored at a population level in distinct age groups. Potential intra-familial, specific effects in adults and children sharing the same socio-economic, cultural level and living habits have been scarcely explored. The investigators aimed to extend the previous observations concerning anthropometric data at the intra-familial level. In particular, The investigators prospectively characterized the variations in lifestyle habits and related outcomes over a 2 two months COVID-19 lockdown period, exploring both parents and their children. A cohort of 149 couple parent/children were prospectively enrolled. By a validated questionnaire The investigators explored changes of Body Mass Index (BMI) and individual lifestyle during a 2-month lockdown.

The pandemic diffusion of the new severe acute respiratory syndrome coronavirus SARS-CoV-2 caused major impacts on health, economy, and social dynamics. During the first wave of the pandemic, besides the direct effect of the COVID-19 disease, staying at home has promoted, in non-infected subjects, sedentary lifestyle, negative psychological consequences, restriction in spending, and accumulation of long-life food with limited use of fresh foods, such as seasonal fruit and vegetables. As a consequence, the lockdown has represented a population-based, inedited model of increased metabolic risk in all age groups, able to affect the health status in a relatively short period.

Previous studies reported negative metabolic outcomes of the lockdown both adults and in children. These effects have been linked with altered eating behavior and lifestyle, with a significant reduction in physical activity, and with an impairment of psychological health. However, these studies were based on self-reported questionnaires, which may lead to misreporting of data. Furthermore, the reported effects on body size variations have been generally explored, at a population level, in separate age groups, and the existence of possible intra-familial, distinct outcomes in adults and children sharing the same critical event and living environment have been scarcely explored.

Although several studies have shown the impact of Lockdown on metabolic status, potential intra-familial, specific effects in adults and children sharing the same socio-economic, cultural level and living habits have been scarcely explored. In the present study The investigators had the chance to dissect the intra-familial impact of two month of lockdown due to COVID-19 pandemic on BMI in a large cohort of non-infected parents and in their children/adolescents.

Primary objective: to characterize changes of dietary habits, lifestyle and anthropometric indices in parents and in their children during lockdown.

The investigators designed an observational, prospective study using a validated questionnaire to profile adults (parents) and their children living in Apulian region (Southern Italy) during the lockdown imposed in the first wave of the pandemic. Overall, 149 parents and 149 children/adolescents are recruited. The study period is 2 months (15 May 2020 - 15 July 2020). Enrolled in the protocol are accompanying parents and children from the outpatient clinics of the Pediatric Unit, in collaboration with the staff of the Unit of Internal Medicine, University of Bari. Participation in the study is on voluntary basis. Children enter the study after parental written informed consent. Adults also provide written informed consent.

Inclusion Criteria:

* Subjects able to sign the Informed Consent
* Subjects who were in Lockdown
* For children, the inclusion criteria were: (i) age between 5 and 18 years; (ii) absence of ongoing therapies.

Exclusion Criteria:

* Subjects not able to provide informed consent
* SARS-CoV-2 infection
* Diagnosis of organic diseases including neoplastic, severe cardiovascular diseases, renal insufficiency, psychiatric disorders.

The investigators considered that a sample of 149 parents and 149 children/adolescents gives sufficient power to detect significant differences over time regarding BMI, physical activity and metabolic status during COVID-19 lockdown

The investigators designed an observational study using a validated questionnaire to profile adults (parents) and their children living in Apulian region (Southern Italy) during the lockdown imposed in the first wave of the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to sign the Informed Consent
* Subjects who were in Lockdown
* For children, the inclusion criteria were: (i) age between 5 and 18 years; (ii) absence of ongoing therapies.

Exclusion Criteria:

* Subjects not able to provide informed consent
* SARS-CoV-2 infection
* Diagnosis of organic diseases including neoplastic, severe cardiovascular diseases, renal insufficiency, psychiatric disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators designed an observational, prospective study using a validated questionnaire to profile adults (parents) and their children living in Apulia region (Southern Italy) during the lockdown imposed in the first wave of the pandemic. Overall, 149 parents and 149 children/adolescents are recruited. The study period is 2 months (15 May 2020 - 15 July 2020). Enrolled in the protocol are accompanying parents and children from the outpatient clinics of the Pediatric Unit, in collaboration with the staff of the Unit of Internal Medicine, University of Bari. Participation in the study is on voluntary basis. Children enter the study after parental written informed consent. Adults also provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Effects of COVID-19 lockdown on changes of anthropometric indices | 2 months
  To characterize changes of dietary habits, lifestyle and anthropometric indices in parents and in their children during lockdown.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanmugam H, Di Ciaula A, Di Palo DM, Molina-Molina E, Garruti G, Faienza MF, vanErpecum K, Portincasa P. Multiplying effects of COVID-19 lockdown on metabolic risk and fatty liver. Eur J Clin Invest. 2021 Jul;51(7):e13597. doi: 10.1111/eci.13597. Epub 2021 May 25. PMID 34032283
- [Background] Di Ciaula A, Krawczyk M, Filipiak KJ, Geier A, Bonfrate L, Portincasa P. Noncommunicable diseases, climate change and iniquities: What COVID-19 has taught us about syndemic. Eur J Clin Invest. 2021 Dec;51(12):e13682. doi: 10.1111/eci.13682. Epub 2021 Sep 29. PMID 34551123
- [Background] Di Renzo L, Gualtieri P, Pivari F, Soldati L, Attina A, Cinelli G, Leggeri C, Caparello G, Barrea L, Scerbo F, Esposito E, De Lorenzo A. Eating habits and lifestyle changes during COVID-19 lockdown: an Italian survey. J Transl Med. 2020 Jun 8;18(1):229. doi: 10.1186/s12967-020-02399-5. PMID 32513197
- [Background] Gornicka M, Drywien ME, Zielinska MA, Hamulka J. Dietary and Lifestyle Changes During COVID-19 and the Subsequent Lockdowns among Polish Adults: A Cross-Sectional Online Survey PLifeCOVID-19 Study. Nutrients. 2020 Aug 3;12(8):2324. doi: 10.3390/nu12082324. PMID 32756458
- [Background] Dunton GF, Do B, Wang SD. Early effects of the COVID-19 pandemic on physical activity and sedentary behavior in children living in the U.S. BMC Public Health. 2020 Sep 4;20(1):1351. doi: 10.1186/s12889-020-09429-3. PMID 32887592
- [Result] Di Renzo L, Gualtieri P, Cinelli G, Bigioni G, Soldati L, Attina A, Bianco FF, Caparello G, Camodeca V, Carrano E, Ferraro S, Giannattasio S, Leggeri C, Rampello T, Lo Presti L, Tarsitano MG, De Lorenzo A. Psychological Aspects and Eating Habits during COVID-19 Home Confinement: Results of EHLC-COVID-19 Italian Online Survey. Nutrients. 2020 Jul 19;12(7):2152. doi: 10.3390/nu12072152. PMID 32707724